CLINICAL TRIAL: NCT07222488
Title: Phase 1/2 Study of Intravesical MK-3120 in BCG-Naïve or BCG-Exposed High-Risk Non-muscle Invasive Bladder Cancer
Brief Title: A Clinical Study of MK-3120 in People With Bladder Cancer (MK-3120-003)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3120-003; U1111-1317-2687 (Registry Identifier: UTN); 2025-520467-40-00 (Registry Identifier: EU CT); MK-3120-003 (Other: MSD)
Record Dates: First submitted 2025-10-27; First posted 2025-10-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Bladder Cancer; Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-3120 (Experimental): Participants will be administered MK-3120 once weekly for the first 6 weeks, followed by once monthly for 9 months.
  Interventions: Biological: MK-3120

INTERVENTIONS:
Biological: MK-3120 — Intravesical administration at one of three doses per protocol
  Other Names: SKB410

SUMMARY:
Researchers are looking for new ways to treat high-risk non-muscle invasive bladder cancer (HR NMIBC). NMIBC is cancer in the tissue that lines the inside of the bladder and has not spread to the bladder muscle or outside of the bladder. In standard treatment for HR NMIBC, doctors first remove the tumor with a procedure called transurethral resection of the bladder tumor (TURBT). Researchers want to learn if using MK-3120, the study medicine, can treat HR NMIBC after TURBT. The goal of this study is to learn about the safety of MK-3120 and if people tolerate it.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed carcinoma in situ (CIS) +/- papillary high-risk non-muscle invasive bladder cancer (NMIBC), confirmed locally.
* Is an individual whose most recent transurethral resection of bladder tumor (TURBT) was performed within 12 weeks before allocation and showed high-risk NMIBC histology. For individuals with papillary tumors (Ta and T1), a complete TURBT must have been performed, as characterized by attainment of a visually complete resection of all papillary tumors (Ta and T1).
* Is either: a) Bacillus Calmette-Guérin (BCG)-naïve, defined as either having never received BCG or having received BCG more than 2 years before CIS +/- papillary high-risk NMIBC recurrence. Recurrence must be at least 24 months from the last exposure to BCG with evidence of complete response during the 2-year period post-BCG OR; b) BCG-exposed and received adequate BCG therapy and had recurrence of CIS +/- papillary high-risk NMIBC >12 months but ≤24 months after the last BCG dose.
* Human immunodeficiency virus (HIV)-infected participants must have well-controlled HIV on antiretroviral therapy.
* Participants who are hepatitis B surface antigen positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to allocation.
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening.

Exclusion Criteria:

* Has history of or current locally advanced (ie, T2, T3, T4) or metastatic urothelial cancer (UC).
* Has concurrent extravesical (ie, urethra, ureter, renal pelvis) non-muscle invasive UC or history of extravesical non-muscle invasive UC that recurred within the last 2 years.
* Has active total bladder incontinence, active urinary tract infection, neurogenic bladder, or urethral stricture.
* Has a condition that would prohibit normal voiding (or holding bladder voiding for 1 to 2 hours).
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, uncontrolled symptomatic arrhythmia, prolongation of QTcF interval to >470 ms, and/or other serious cardiovascular and cerebrovascular diseases within the 6 months preceding study intervention.
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has active infection requiring systemic therapy.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease (ILD) that required steroids, or has current pneumonitis/ILD.
* Has not adequately recovered from major surgery or has ongoing surgical complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Dose-limiting Toxicity (DLT) | Up to approximately 5 weeks
  Any of the following toxicities will be considered a DLT:
  Hematuria leading to clot or obstruction; Grade (Gr) 4 thrombocytopenia; Gr 3 thrombocytopenia associated with clinically significant bleeding; Febrile neutropenia for more than 1 hour; Other Gr ≥3 hematologic toxicity lasting >7 days; Nonhematologic AE ≥Gr 3 (with exceptions); ≥Gr 2 pneumonitis/ interstitial lung disease; Any ≥Gr 3 nonhematologic laboratory value if clinically significant medical intervention is required, leads to hospitalization, persists for >7 days, results in a drug induced liver injury, or elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) lab value >8 ×upper limit of normal (ULN) regardless of duration and AST or ALT elevation 5 × to 8 × ULN that persists for greater than 2 weeks; Recurrent Gr 2 AE resulting in >2 weeks delay in receiving the next treatment dose; Any intervention-related toxicity that results in study intervention discontinuation; Gr 5 toxicity or AE.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 24 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Number of Participants Who Discontinue Study Treatment Due to AEs | Up to approximately 12 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | Up to approximately 3 months
  CR is defined as the absence of all of the following as determined by local assessment using urine cytology, cystoscopy, biopsy and radiology assessments as applicable:
  * High-risk non-muscle invasive urothelial cancer (UC) (defined as high-grade [HG] noninvasive papillary [Ta], carcinoma in situ [CIS], or any submucosal invasive [T1] disease of the bladder, urethra, or upper tract [ureters, renal pelvis])
  * Any muscle invasive tumor (T2) or greater in the bladder, including transurethral prostate stromal invasion of UC, or in the upper tract (ureters, renal pelvis)
  * Metastatic UC, defined as:
    * Regional lymph node metastasis of UC (N1 or greater)
    * Distant lymph node or visceral metastasis of UC (M1)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- United States (2):
  - Michael G Oefelein Clinical Trials ( Site 0005), Bakersfield, California
  - Carolina Urologic Research Center ( Site 0006), Myrtle Beach, South Carolina
- CHU de Quebec - Hopital de l'Enfant-Jesus ( Site 0011), Québec, Quebec, Canada
- Rabin Medical Center ( Site 0062), Petah Tikva, Israel
- Ankara University Health Practice and Research Hospitals ( Site 0132), Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/